CLINICAL TRIAL: NCT05300802
Title: The Role of Dexmedetomidine As Myocardial Protection In Pediatric Cyanotic Congenital Heart Disease Undergoing Open Cardiac Surgery Using Cardiopulmonary Bypass Machine: A Preliminary Study
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Cardiovascular Center Harapan Kita Hospital Indonesia (Other)
Responsible Party: Principal Investigator, Dian Kesumarini, MD, Principal Investigator, National Cardiovascular Center Harapan Kita Hospital Indonesia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LB.02.01/VII/581/KEP058/2021; LB.02.01/VII/581/KEP058/2021 (Other: National Cardiovascular Center Harapan Kita Hospital Indonesia)
Record Dates: First submitted 2021-12-20; First posted 2022-03-29 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Congenital Heart Disease in Children; Cardiopulmonary Bypass
Keywords: Dexmedetomidine; Myocardial Protection; Pediatric Cyanotic Congenital Heart Disease; Cardiopulmonary Bypass; Aristotle Score
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Placebo Comparator): Ringer acetate
  Interventions: Drug: Placebo
- Group B (Experimental): Priming Dexmedetomidine 1 mcg/kg, Intravenous Ringer acetate
  Interventions: Drug: Dexmedetomidine Hcl 100 Mcg/mL Inj
- Group C (Experimental): Priming Dexmedetomidine 0.5 mcg/kg, Intravenous Dexmedetomidine 0.25 mcg/kg/hour
  Interventions: Drug: Dexmedetomidine Hcl 100 Mcg/mL Inj

INTERVENTIONS:
Drug: Placebo — 50 ml of Ringer acetate will be added to the priming solution and followed by a continuous 50 ml infusion of Ringer acetate running at 25 ml/hour.
  Other Names: Ringer Acetate
  Arms: Group A
Drug: Dexmedetomidine Hcl 100 Mcg/mL Inj — 1 mcg/kg diluted DEX will be added to the priming solution and followed by a continuous infusion of 50 ml Ringer acetate running at 25 ml/hour.
  Other Names: Kabimidine
  Arms: Group B
Drug: Dexmedetomidine Hcl 100 Mcg/mL Inj — 0.5 mcg/kg DEX will be added to the priming solution and followed by a continuous infusion of 0.25 mcg/kg/hour DEX diluted in 50 ml of ringer acetate running at 25 ml/hour.
  Other Names: Kabimidine
  Arms: Group C

SUMMARY:
Congenital Heart Diseases (CHD) are one of the most common congenital anomalies. Worldwide, 8 to 9 out of 1000 of children are born with a CHD, of which 25 percent of are cyanotic CHD. In Indonesia, the prevalence is 43.200 out of 4.8 million births annually. The morbidity and mortality of cyanotic CHDs in the National Cardiovascular Center Harapan Kita (NCCHK) are higher than acyanotic CHDs. Open-heart surgery using a cardiopulmonary bypass (CPB) machine temporarily takes over the function of the heart and lung during surgery. However, the use of CPB has several negative effects such myocardial injury, systemic inflammation, and reperfusion injury. Preoperative hypoxia in cyanotic CHD tends to be associated with a higher risk of myocardial injury. Myocardial protection has an important role in attenuating those effects. Generally, we use a cardioplegia solution as myocardial protection, but there are several non-cardioplegia techniques that can be used to enhance myocardial protection during cardiac bypass, such as adding an anesthetic agent. Dexmedetomidine (DEX) is the active dextroisomer of medetomidine, a selective α-2 adrenergic, which has major effects including hypnosis, sedation, and analgesia as well as cardiovascular effects. The sedation is induced by stimulating the α-2 adrenergic receptor in the locus coeruleus (LC) in the pons cerebri. DEX also increases the level of GABA and Galanin and reduces endogenous norepinephrine. The lower level of endogenous norepinephrine decreases the afterload of the ventricles, increases cardiac output, and reduces myocardial injury as a result. Furthermore, the peripheral effects of DEX can reduce myocardial ischemia-reperfusion (MIR) by inhibiting NF-кB pathway activation and reducing the number of proinflammatory cytokines released. Research related to the priming and infusion of DEX during CPB in patients with cyanotic CHDs who are undergoing open-heart surgery is less reported. The aims of this study are to determine the effectiveness of the priming and infusion of DEX during CPB as myocardial protection by using two different doses compared to the control group. The population included in this study is pediatric patients with cyanotic CHD who are undergoing open-heart surgery using CPB and who classified as 6 to 9 in the Aristotle Score.

DETAILED DESCRIPTION:
The investigators will conduct a double-blind randomized controlled trial preliminary study to determine the effectiveness of the priming and infusion of DEX during CPB as myocardial protection by using two different doses compared to the control group. The population included in this study will be pediatric patients with cyanotic CHD who are undergoing open-heart surgery using CPB and who classified as 6 to 9 in the Aristotle Score. This study was approved by the research ethical committee (Institutional Review Board) of the National Cardiovascular Center Harapan Kita Jakarta (NCCHK). Before randomization, participants who are eligible based on inclusion and exclusion criterias will be given informed consent. If the guardians of the patients agree, the patient will be included in this research. Fifteen pediatric patients with cyanotic CHD will be randomly divided into three groups A, B, and C. Group A is the control group and will be given 50 ml Ringer acetate solution in a 50 ml syringe that will be added to the priming solution in CPB, followed by 50 ml of Ringer acetate solution administered in a syringe pump infusion running at 25 ml/hour and which will be ended by the end of CPB. Group B will received DEX 1 mcg/kg diluted in 50 ml of Ringer acetate solution in a 50 ml syringe added in the priming solution in CPB, followed by 50 ml of Ringer acetate solution administered in a syringe pump infusion running at 25 ml/hour and which will be ended by the end of CPB. Group C will be administered 0.5 mcg/kg DEX, diluted in 50 ml of Ringer acetate solution in a 50 ml syringe added in the priming solution in CPB, followed by 0.25 mcg/kg/hour DEX diluted in 50 ml of Ringer acetate solution administered in a syringe pump infusion running at 25 ml/hour infusion which will be ended by the end of CPB.

Age, gender, body weight, body length, body surface area, Aristotle scores, aortic cross-clamp time, CPB time, and operation time are included as demographics and characteristics data. The investigators will measure myocardial injury biomarker serum levels (Troponin I) and cytokines proinflammatory biomarker serum levels (IL-6) as the primary outcome of myocardial protection. Serum levels of troponin I and IL-6 will be taken 4 times (T1: 5 minutes after induction as baseline level; T2: 1 hour after CPB; T3: 6 hours after CPB, and T4: 24 hours after CPB). Secondary outcomes include hemodynamic profile (Cardiac output, cardiac index, and systemic vascular resistance, at 6 hours, 24 hours, and 48 hours after CPB plus serum lactate levels at 5 minutes after induction as baseline level, 1 hour, 6 hours, and 24 hours after CPB), morbidity outcomes (the highest Vasoinotropic Score at the first 24 hours after CPB, length of mechanical ventilation, and length of intensive care stay), and adverse event occurrences such as hypotension and bradycardia (at 5 minutes after induction as baseline level, 1 hour, 6 hours, and 24 hours after CPB).

ELIGIBILITY:
Inclusion Criteria:

* All the patients guardian consent to participate in this study
* Patient with Cyanotic CHD who are undergoing open-heart surgery using CPB with an Aristotle score of 6-9
* Patient is aged between 1 month to 6 years

Exclusion Criteria:

* Elective surgery patients who change into an emergency case surgery
* Patient with procalcitonin levels exceeding 0.5 ng/ml with the symptoms of infection
* Patient with liver dysfunction as measured by an increase of Glutamic Oxaloacetic Transaminase (SGOT)/ Serum Glutamic Pyruvic Transaminase (SGPT) levels more than 1.5 times from baseline
* Patient with Renal dysfunction as measured by creatinine levels exceeding 2 mg/dL

Drop out Criteria:

* Duration of CPB and/or Aortic cross-clamp time exceeding 120 minutes
* Intraoperative anatomy of CHDs finding is different from the preoperative diagnosis so that the patient no longer fulfils the Aristotle score of 6-9
* Surgery requires more than two attempts of CPB
* Patient fails to wean from CPB
* Patient requires ECMO (Extracorporeal Membrane Oxygenator) postoperatively
* Patient dies on the operating table

Ages: 1 Month to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-07-16 (Actual)

PRIMARY OUTCOMES:
Serum Troponin I at baseline | 5 minutes after induction of anesthesia (T1)
  Troponin I serum concentration will be measured using RnD Quantikine reagent (ng/mL)
Serum Troponin I at 1 hour after cardiopulmonary bypass | 1 hour after cardiopulmonary bypass (T2)
  Troponin I serum concentration will be measured using RnD Quantikine reagent (ng/mL)
Serum Troponin I at 6 hours after cardiopulmonary bypass | 6 hours after cardiopulmonary bypass (T3)
  Troponin I serum concentration will be measured using RnD Quantikine reagent (ng/mL)
Serum Troponin I at 24 hours after cardiopulmonary bypass | 24 hours after cardiopulmonary bypass (T4)
  Troponin I serum concentration will be measured using RnD Quantikine reagent (ng/mL)
Serum IL-6 at baseline | 5 minutes after induction of anesthesia (T1)
  IL-6 serum concentration will measured using an Elecsys IL-6 reagent (pg/mL)
Serum IL-6 at 1 hour after cardiopulmonary bypass | 1 hour after cardiopulmonary bypass (T2)
  IL-6 serum concentration will measured using an Elecsys IL-6 reagent (pg/mL)
Serum IL-6 at 6 hours after cardiopulmonary bypass | 6 hours after cardiopulmonary bypass (T3)
  IL-6 serum concentration will measured using an Elecsys IL-6 reagent (pg/mL)
Serum IL-6 at 24 hours after cardiopulmonary bypass | 24 hours after cardiopulmonary bypass (T4)
  IL-6 serum concentration will measured using an Elecsys IL-6 reagent (pg/mL)

SECONDARY OUTCOMES:
Cardiac output | 6 hours (T3), 24 hours (T4), and 48 hours (T5) after cardiopulmonary bypass
  Cardiac output will be measured using transthoracic echocardiography (L/min)
Cardiac Index | 6 hours (T3), 24 hours (T4), and 48 hours (T5) after cardiopulmonary bypass
  Cardiac index will be measured using transthoracic echocardiography (L/min)
Systemic Vascular Resistance (SVR) | 6 hours (T3), 24 hours (T4), and 48 hours (T5) after cardiopulmonary bypass
  SVR will be measured using transthoracic echocardiography (L/min)
Serum Lactate | 5 minutes after anesthesia induction (T1), and then 1 hour (T2), 6 hours (T3), and 24 hours (T4) after cardiopulmonary bypass
  Serum lactate will be measured using an enzymatic method with a blood gas analyzer machine (mmol/L)
VIS Score | 6 hours (T3), 24 hours (T4), and 48 hours (T5) after cardiopulmonary bypass
  Vasoinotropic score will be measured using the VIS formula
Mechanical ventilation time | 3 days (or until the patient is extubated)
  Mechanical ventilation time will be measured from the moment the patient arrives at the intensive care unit until the patient is extubated
Hospital length of stay in the intensive care unit | 7 days (or until the patient is discharge from intensive care unit)
  Hospital length of stay in the intensive care unit will be measured from the moment the patient is admitted to the intensive care unit after the surgery until discharge from intensive care unit
Adverse effects of DEX related to the hemodynamic profile ( hypotension and bradycardia) | 5 minutes after anesthesia induction (T1), and then 1 hour (T2), 6 hours (T3), 24 hours (T4), and 48 hours (T5) after cardiopulmonary bypass
  Adverse effects of DEX related to the hemodynamic profile ( hypotension and bradycardia)

CONTACTS AND LOCATIONS:
Locations (1):
- National Cardiovascular Center Harapan Kita Hospital Indonesia, Jakarta, Indonesia